CLINICAL TRIAL: NCT05584878
Title: Clinical and Topographic Evaluation of the Remineralizing Potential of Biomimetic Scaffolds on Enamel White Spot Lesions (a Randomized Controlled Clinical Trial and In-vitro Study)
Brief Title: Remineralizing Potential of Biomimetic Scaffolds on Enamel White Spot Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: biomimetic scaffolds _2022
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: White Spot Lesion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental)
  Interventions: Other: Curodont repair Self- assembling peptide P11-4
- Group II (Experimental)
  Interventions: Other: Ph-chi phosphorylated - nano-chitosan
- Group III (Active Comparator)
  Interventions: Other: CCP-ACP " +ve control " Casein phosphopeptide amorphous calcium phosphate

INTERVENTIONS:
Other: Curodont repair Self- assembling peptide P11-4 — The labial surface of each tooth in both arches from central to the first premolar on both sides will be treated by Curodont
  Arms: Group I
Other: Ph-chi phosphorylated - nano-chitosan — The labial surface of each tooth in both arches from central to the first premolar on both sides will be treated by Ph-chi phosphorylated - nano-chitosan
  Arms: Group II
Other: CCP-ACP " +ve control " Casein phosphopeptide amorphous calcium phosphate — The labial surface of each tooth in both arches from central to the first premolar on both sides will be treated by CCP-ACP
  Arms: Group III

SUMMARY:
The modern concept in caries treatment focuses on the non-invasive approach and on the biomimetic remineralization of early non-cavitated white spot carious lesions. Recently developed biomimetic scaffolds attempt to remineralize the dental tissues and are more regenerative than reparative.

ELIGIBILITY:
Inclusion Criteria:

* Patients who at least have 1 white spot lesion.
* No systemic diseases or taking any medication affecting salivary flow.
* Patients with good oral hygiene measures.
* Patients with moderate caries risk assessment.
* Post orthodontic WSLs with International Caries Detection and Assessment System (ICDAS II) scoring criteria (1-2).

Exclusion Criteria:

* Participant in another trial.
* Developmental non carious lesion (enamel hypoplasia and dental fluorosis).
* Presence of abnormal oral disease, or medically compromised patients.
* Participants who had evidence of reduced salivary flow or significant tooth wear.
* Allergy to milk products or other drug allergies.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in DIAGNOdent values | Baseline, 1 month, 3 months , 6 months, 9 months, 12 months
  The DIAGNOdent uses laser fluorescence to aid in the detection of caries within the tooth structure.
change in ICDAS scores | Baseline, 1 month, 3 months , 6 months, 9 months, 12 months
  Code Description 0: Sound tooth surface: No evidence of caries after 5 sec air drying
  1. First visual change in enamel: Opacity or discoloration (white or brown) is visible at the entrance to the pit or fissure seen after prolonged air drying
  2. Distinct visual change in enamel visible when wet, lesion must be visible when dry
  3. Localized enamel breakdown (without clinical visual signs of dentinal involvement) seen when wet and after prolonged drying
  4. Underlying dark shadow from dentine
  5. Distinct cavity with visible dentine
  6. Extensive (more than half the surface) distinct cavity with visible dentine

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Soliman EM, Abdelfattah WM, Mohamed DR, Nagui DA, Holiel AA. Clinical evaluation of the remineralizing potential of biomimetic scaffolds on enamel white spot lesions: A 12-month randomized controlled trial. J Dent. 2025 Dec 16;166:106303. doi: 10.1016/j.jdent.2025.106303. Online ahead of print. PMID 41412271